CLINICAL TRIAL: NCT00725179
Title: Treatment of Acetaminophen Toxicity With Intravenous vs Oral N-acetylcysteine: A Retrospective Review
Brief Title: Treatment of Acetaminophen Toxicity With N-acetylcysteine
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Martha Blackford, PharmD, Akron Children's Hospital
Other Study IDs: APAP & NAC
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Acetaminophen Toxicity
Keywords: acetaminophen toxicity; n-acetylcysteine; liver toxicity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients receiving oral NAC treatment
- 2: Patients receiving IV NAC treatment

SUMMARY:
Retrospective chart review of patients who received N-acetylcysteine for APAP toxicity to assess length of oral vs IV treatment and overall healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to CHMCA between June 1, 2004 to May 31, 2008 with a qualifying ICD-9 diagnosis code for the following APAP overdose situations; poisoning, accidental, suicide attempt, therapeutic use, assault, and undetermined (965.4, E850.4, E950.0, E935.4, E962.0, E980.0)
* Serum APAP concentrations ≥ 150 g/mL at 4 hours or a serum concentration above the possible hepatotoxic line on the Rumack-Matthew's nomogram if obtained > 4 hours post ingestion
* Between the ages of 0-21 years

Exclusion Criteria:

* Serum APAP concentrations are not actually documented
* Patient did not receive oral or IV NAC treatment
* Patient has a preexisting liver disease such as cirrhosis or hepatitis C
* Patient > 21 years of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adolescent patients with acetaminophen toxicity
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Duration of oral vs IV NAC treatment in hours | From admission to discharge

SECONDARY OUTCOMES:
Overall healthcare costs associated with IV vs Oral NAC treatment | From admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Martha Blackford, PharmD, Principal Investigator — CHMCA
Locations (1):
- Children's Hospital Medical Center of Akron, Akron, Ohio, United States

REFERENCES:
- [Background] Heard KJ. Acetylcysteine for acetaminophen poisoning. N Engl J Med. 2008 Jul 17;359(3):285-92. doi: 10.1056/NEJMct0708278. PMID 18635433
- [Background] Culley CM, Krenzelok EP. A clinical and pharmacoeconomic justification for intravenous acetylcysteine: a US perspective. Toxicol Rev. 2005;24(2):131-43. doi: 10.2165/00139709-200524020-00007. PMID 16180933
- [Background] Kanter MZ. Comparison of oral and i.v. acetylcysteine in the treatment of acetaminophen poisoning. Am J Health Syst Pharm. 2006 Oct 1;63(19):1821-7. doi: 10.2146/ajhp060050. PMID 16990628
- [Derived] Blackford MG, Felter T, Gothard MD, Reed MD. Assessment of the clinical use of intravenous and oral N-acetylcysteine in the treatment of acute acetaminophen poisoning in children: a retrospective review. Clin Ther. 2011 Sep;33(9):1322-30. doi: 10.1016/j.clinthera.2011.08.005. Epub 2011 Sep 3. PMID 21890206